CLINICAL TRIAL: NCT01217320
Title: Efficacy and Safety of Creatine Supplementation in Patients With Juvenile Systemic Lupus Erythematosus and Juvenile Dermatomyositis
Brief Title: Creatine Supplementation in Pediatric Rheumatology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cr in rheumato
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Juvenile Systemic Lupus Erythematosus; Juvenile Dermatomyositis
Keywords: rheumatology; creatine supplementation; quality of life; strength; juvenile systemic lupus erythematosus; juvenile dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — Creatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- creatine supplementation (Experimental): will receive 5g/d of creatine monohydrate throughout the trial
  Interventions: Dietary Supplement: creatine
- placebo (Placebo Comparator): will receive 5g/d of placebo (dextrose) throughout the trial
  Interventions: Dietary Supplement: placebo (dextrose)

INTERVENTIONS:
Dietary Supplement: creatine — 5g/d throughout 12 weeks
  Arms: creatine supplementation
Dietary Supplement: placebo (dextrose) — 5g/d throughout 12 weeks
  Arms: placebo

SUMMARY:
Creatine supplementation may improve strength, muscle mass, bone mass and muscle function in healthy and elderly people. The investigators speculate that creatine supplementation could have therapeutic effects in pediatric rheumatic (i.e., juvenile systemic lupus erythematosus and juvenile dermatomyositis) patients who usually present muscle weakness, muscle wasting and bone mass loss.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with lupus systemic erythematosus and juvenile dermatomyositis
* physically inactive
* stable pharmacological treatment

Exclusion Criteria:

* macroalbuminuria
* GFR < 30 mL/min/1.73m2
* use of oral anticontraceptive agents
* pregnancy
* diabetes mellitus
* hypothyroidism

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
muscle strength | after six months

SECONDARY OUTCOMES:
kidney function parameters | after six months
quality of life | after six months
muscle function | after six months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD, Study Director — University of Sao Paulo; Eloisa Bonfa, MD, PhD, Study Director — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Hayashi AP, Solis MY, Sapienza MT, Otaduy MC, de Sa Pinto AL, Silva CA, Sallum AM, Pereira RM, Gualano B. Efficacy and safety of creatine supplementation in childhood-onset systemic lupus erythematosus: a randomized, double-blind, placebo-controlled, crossover trial. Lupus. 2014 Dec;23(14):1500-11. doi: 10.1177/0961203314546017. Epub 2014 Aug 18. PMID 25135060